CLINICAL TRIAL: NCT07172490
Title: Interdisciplinary Program to Improve the Lifestyle of People With Complex Chronic Pathologies in the Alt Pirineu and Aran Region Using the APA-FIT App: Randomized Controllled Trial.
Brief Title: Interdisciplinary Program to Improve Lifestyle in Chronic Pathology: Alt Pirineu Aran in Fit (APA-FIT)
Acronym: APA-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: CatSalut Catalonia, Spain (Unknown)
Responsible Party: Principal Investigator, Marta Prats Arimon, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDIAP JORDI GOL 24/163-ACps
Record Dates: First submitted 2025-08-25; First posted 2025-09-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Non-communicable Diseases (NCD); Cardiovascular Risk; Obesity Prevention
Keywords: Physical Activity; Nutrition; Mental Health; Digital Tools
MeSH Terms: conditions — Noncommunicable Diseases; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A multicenter, quasi-experimental pre-post study with two parallel arms-intervention group (IG) and control group (CG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) Normal healthcare (No Intervention): 1. Moderate cardiovascular risk: Standard physical-activity and nutrition counseling
     • Assessments: Identical to Branch 1 for nutrition, bioimpedance, PA, and fitness test
  2. High cardiovascular risk: Standard physical-activity and nutrition counseling. • Assessments: Identical to Branch 2 for nutrition, bioimpedance, PA, and fitness test
- Intervention Group (IG) APP digital tool (Experimental): 1. Moderate cardiovascular Risk
     . Assessments: Identical to Branch 1 for nutrition, anthropometry/bioimpedance, PA, and fitness
     • Risk Monitoring: ECG (if none performed in last six months) and blood tests at the reference primary-care clinic
  2. High cardiovascular risk
     * Assessments: Nutritional habits; anthropometry and/or bioimpedance; habitual PA evaluation; fitness testing
     * Risk Monitoring: Fasting blood assays and risk-factor management at participants' primary care clinic
     * Exercise Testing: Maximal exercise tests with gas analysis
       * At Hospital de Cerdanya's Sports Medicine Unit for patients from Puigcerdà and la Seu d'Urgell-Oliana
       * Mobile Sports Medicine teams (portable gas analyzers, laptop, cycle ergometer) for remaining sites
       * All tests supervised by a sports cardiologist
  Interventions: Other: APA-FIT interdisciplinary program

INTERVENTIONS:
Other: APA-FIT interdisciplinary program — Intervention: APA-FIT
  The APA-FIT program is an interdisciplinary intervention targeting three core domains in adults with chronic conditions at moderate or high risk for physical activity (PA): physical exercise, nutritional habits, and positive mental health. Over nine months, participants receive:
  * Individualized PA Prescription
    * Bimonthly follow-up visits with a certified PA prescriber (physician, nurse, or physiotherapist)
    * Weekly supervised exercise sessions led by a coach
    * Automated PA logging and goal tracking via the APA-FIT app
  * Nutritional Counseling
    * Initial and final dietary assessments with a registered nutritionist
    * Bimonthly follow-up and three hands-on Mediterranean-diet workshops
  * Psychosocial Support for Positive Mental Health
    * Four bimonthly group sessions facilitated by the primary-care emotional-well-being lead
    * In-app materials, peer support features, and one-on-one check-ins
  Arms: Intervention Group (IG) APP digital tool

SUMMARY:
Interdisciplinary Program to Improve the Lifestyle of Individuals with Chronic Conditions in the Alt Pirineu and Aran Region

Sedentary behavior and lack of regular physical activity have been widely recognized as urgent global public health issues-not only because they are key risk factors for cardiovascular morbidity and mortality, but also due to their impact on major chronic diseases.

Primary Objective / Hypothesis To evaluate the effectiveness of an intervention program aimed at improving the lifestyle of individuals with chronic conditions in the Alt Pirineu and Aran health region by promoting active living and physical activity (PA), healthy dietary habits, and positive mental health (PMH), through the use of a digital tool (APP). The program also aims to determine whether this intervention leads to a reduction in cardiovascular risk, comorbidity, and premature aging associated with non-communicable diseases.

Study Design and Sample The sample will consist of individuals over 18 years of age with moderate to high cardiovascular risk who voluntarily participate in the project. The program will last for 9 months and will be structured into two groups: an intervention group, which will actively participate in the program through the APP, and a control group, which will not receive the intervention. Pre- and post-intervention measurements will be applied to assess the effects of the program.

Applicability and Relevance This project seeks to implement an interdisciplinary care model for individuals with chronic conditions, aiming to enhance lifestyle behaviors, reduce comorbidity, and mitigate premature aging. The APA-fit digital tool seeks to implement this model by empowering patients in their self-care and facilitating seamless, effective communication between patients and healthcare professionals.

DETAILED DESCRIPTION:
Project Justification: Lifestyle, Physical Activity and Public Health

A sedentary lifestyle and lack of regular physical activity have been widely recognised as major global public health concerns. These behaviours are not only significant risk factors for cardiovascular morbidity and mortality, but are also strongly associated with the development and progression of chronic diseases such as cancer, obesity, and type 2 diabetes mellitus. According to the World Health Organization (WHO), physical inactivity accounts for 25% of breast and colon cancer cases, 27% of diabetes cases, and 30% of ischaemic heart disease cases. These figures underscore the urgent need for preventive and therapeutic interventions focused on promoting physical activity and healthy lifestyle habits.

Globally, the prevalence of sedentary behaviour is estimated at 49.7%. A person is considered sedentary if they spend more than five hours seated per day and engage in less than 90 minutes of physical activity per week. Physical activity is defined as any bodily movement produced by skeletal muscles that results in a substantial increase in energy expenditure. This includes everyday activities such as walking, climbing stairs, performing household chores, or shopping. In contrast, exercise refers to planned, structured, and repetitive physical activity aimed at improving or maintaining physical fitness, health, and quality of life. The American College of Sports Medicine (ACSM) recommends that adults engage in moderate-intensity exercise for at least 30 minutes per day, five days per week, or vigorous-intensity exercise for 20 minutes per day, three days per week.

Concurrently, dietary habits have deteriorated, particularly in developed countries, due to accelerated lifestyles, irregular meal patterns, and the widespread availability of ultra-processed foods. These changes have led to increased consumption of products high in sugars, saturated fats, and salt, and a decline in the intake of foods associated with healthy dietary patterns, such as the Mediterranean diet. This diet is characterised by a high intake of fruits, vegetables, legumes, nuts, whole grains, fish, and extra virgin olive oil, and a low intake of red and processed meats. The PREDIMED study has demonstrated that adherence to the Mediterranean diet significantly reduces the risk of cardiovascular events such as acute myocardial infarction and stroke.

The combination of sedentary behaviour and poor dietary habits has contributed to a sustained rise in obesity prevalence, which has become one of the leading public health challenges. The WHO defines obesity as an abnormal or excessive accumulation of body fat that may impair health. It is diagnosed when the body mass index (BMI) is equal to or greater than 30 kg/m². In women, obesity is defined by a body fat percentage exceeding 35%, and in men, 30%. In Spain, the National Health Survey (2015) reported that 53.7% of adults were overweight or obese, and among children and adolescents (aged 2 to 17), the prevalence reached 27.8%. In Catalonia, the 2020 Health Survey indicated that 20% of the adult population was sedentary, rising to 38.1% when minimally active individuals were included. Furthermore, 33.7% of individuals over the age of 15 were overweight, and 17% were obese, with a clear upward trend.

Scientific literature has also established a link between obesity, sedentary behaviour, and psycho-emotional disorders such as depression and anxiety. These conditions may act both as risk factors and consequences of unhealthy lifestyles, creating a vicious cycle that is difficult to break. Several studies have shown that multidisciplinary interventions combining physical exercise, nutritional education, and behavioural support can significantly improve the physical and emotional health of individuals with obesity, reducing comorbidities and the need for pharmacological or invasive treatments such as bariatric surgery.

There is robust scientific evidence supporting the benefits of regular moderate physical activity and healthy eating habits. Physically, these practices help reduce the risk of cardiovascular disease, hypertension, type 2 diabetes, and other metabolic disorders. Psychologically, they promote autonomy, self-esteem, regulation of sleep-wake cycles, and a reduction in anxiety and depression symptoms.

In response to this public health challenge, various initiatives and intervention programmes have been developed at international, national, and regional levels. At the European level, the EUPAP (European Physical Activity on Prescription) programme, led by the Swedish Public Health Agency and the Swedish Association of Physical Activity Professionals, promotes physical activity prescription as a tool to improve health, prevent non-communicable diseases, and reduce health inequalities. The Swedish model is currently being adapted and implemented in several European regions, including Catalonia, where the *Caminem* project has been active since 2012.

In Spain, the NAOS Strategy (Nutrition, Physical Activity and Obesity Prevention) promotes physical activity in schools, educational institutions, and workplaces, as well as a balanced diet based on the Mediterranean pattern. In Catalonia, the PAAS (Comprehensive Plan for the Promotion of Health through Physical Activity and Healthy Eating), developed by the Department of Health, coordinates actions across five domains: education, healthcare, community, workplace, and communication. This plan aligns with the WHO's global strategy and the NAOS framework established by the Spanish Agency for Consumer Affairs, Food Safety and Nutrition.

This context highlights the need to develop and evaluate new interdisciplinary intervention programmes that integrate physical activity, nutritional education, and emotional support as central components for health promotion and chronic disease prevention. These programmes must be adaptable to diverse contexts and population groups, particularly in regions with specific geographical and socioeconomic characteristics, such as mountainous or rural areas.

The proposed project is framed within this strategic approach and aims to improve the health and quality of life of the population by promoting an active and healthy lifestyle. Through a structured, evidence-based intervention, the project seeks to reduce the prevalence of sedentary behaviour, obesity, and associated disorders, while enhancing emotional well-being and social cohesion. Rigorous evaluation of outcomes will generate transferable knowledge and contribute to the development of more effective and sustainable public health policies.

Methodology

This study employs a two-phase quantitative design:

1. Phase I: A cross-sectional, descriptive observational study of a sample of 520 participants.
2. Phase II: A randomized controlled trial with two arms (intervention vs. control), stratified by high versus moderate cardiovascular risk, using a pre-post test model.

The study will be conducted across eight primary care areas in the Alt Pirineu and Aran region, with sample sizes allocated according to local population density. The nine-month interdisciplinary intervention comprises three core strategies:

* Physical Activity Prescription
* Healthy Nutritional Habits
* Positive Mental Health

Monitoring and follow-up will be performed via the APA-fit app-web platform. Assessment tools include:

* Physical Activity & Fitness: International Physical Activity Questionnaire; Rapid Physical Activity Classifier; 6-minute walk test; graded exercise test
* Nutrition: Mediterranean Diet Adherence Screener; Food Frequency Questionnaire
* Body Composition & Metabolic/Cardiovascular Risk: Advanced anthropometry; bioelectrical impedance analysis
* Psychosocial Health: Positive Mental Health Questionnaire
* General Health: Lipid and glucose blood profile; evaluation of toxic habits; clinical history

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, diagnosed with one or more chronic conditions
* Classified as having moderate or high cardiovascular risk for physical activity Moderate Risk: Men ≥ 45 and women ≥ 55 years. Two or more cardiovascular (CV) risk factors High Risk: One or more signs or symptoms of cardiovascular, respiratory, or metabolic disease.Diagnosed cardiovascular or metabolic disease
* Referred by a primary care physician or community nurse who deems a lifestyle change necessary to improve health and quality of life
* Ownership of a smartphone with internet access, camera capability, and sufficient internal storage to install and run the APA-FIT app Participants meeting these criteria will be invited to enroll in the study and randomized to either the intervention or control arm for the Phase II evaluation. Continuous monitoring and follow-up will occur throughout the nine-month program and at 3- and 6-month post-intervention checkpoints.

Exclusion Criteria:

* [Not provided; assume standard medical or logistical exclusions will apply.]

Exclusion Criteria Phase II

1. Severe visual or hearing impairments that would preclude participation in the intervention
2. Significant cognitive disorders
3. Dependence in activities of daily living
4. Failure to adhere to the therapeutic commitment and/or provide informed consent
5. Any medical condition that contraindicates physical activity or otherwise prevents completion of the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 520 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of frecuency and intensity of pysical activity | From enrollment to end of treatment , 9 months
  The CLASS-AF (Quick Physical Activity Rating Scale) is a brief tool to estimate habitual physical activity without lengthy questionnaires. It assesses four core items: weekly frequency of moderate/vigorous activity (0-4 pts), average duration per session (0-4 pts), perceived intensity (light = 1, moderate = 2, vigorous = 3 pts), and leisure-time activity level (0-3 pts). Scores are summed (range 0-14) to classify activity: low/sedentary (0-4), moderate (5-9), or high (10-14).
Change from baseline mediterrainian diet on 14 points on the scale of adherence to the Mediterranean diet. | from enrollment to end the treatment. 9 months
  Description: The scale of adherence to the Mediterranean diet, is a scale based on 14 items where you ask about 7 groups of foods and portions characteristic of this diet. each item must score with a 1 or 0 depending on the fulfilled or not. The sum of the points if it is less than 9 indicates a bad grip if it is equal to or greater than 9 , a good grip
Change from baseline of positive mental health based on 18 points of the Positive Mental Health Scale-Revised | From enrollment to end the treatment. 9 months
  Change from baseline of positive mental health based on 18 points of the Positive Mental Health Scale-Revised Description: The SMP multifactorial scale revised, consists of 18 items that are distributed among 6 factors: Personal Satisfaction, Prosocial Attitude, Self-Control, Autonomy, Problem Solving and Self-Update, and Interpersonal Relationship Skills. The evaluation of each item is done with a scale scale ranging from 1 to 4. Being 1, always or almost always, 2, quite often, 3 often and 4, never or almost never. Finally, a score between 18 and 72 is obtained, the higher the score the more positive mental health.
Change from baseline of the BMI of participants. Weight and height will be combined to report BMI in kg/m^2 | From enrollment to end of treatment, 9 months
  The formula (weight/height m²) will be applied to measure Body Mass Index (BMI).
Height of participants | baseline
  The height will be measured with a measuring tape in meters. Participants will be measured without shoes.
Change from baseline of the weight of participants | From enrollment to end of treatment, 9 months
  Weigh will be mesured with a analogic weighing machine in Kilograms. Participants are mesured only with underwear clouths
Change from baseline of water percentage with a bioimpedance scale | From enrollment and each 3 month (3, 6, 9)
  Participants are measured only with underwear cloths on the bioimpedance scale TANITA BC 602
Change from baseline of fat mass percentage and kg with a bioimpedance scale | From enrollment and each 3 month (3, 6, 9)
  Participants are measured only with underwear cloths on the bioimpedance scale TANITA BC 602
Change from baseline of muscle percentage and kg with a bioimpedance scale | From enrollment and each 3 month (3, 6, 9)
  Participants are measured only with underwear cloths on the bioimpedance scale TANITA BC 602
Change from baseline of bone percentage and kg with a bioimpedance scale | From enrollment and each 3 month (3, 6, 9)
  Participants are measured only with underwear cloths on the bioimpedance scale TANITA BC 602
Change from baseline of fat free mass percentage and kg with a bioimpedance scale | From enrollment and each 3 month (3, 6, 9)
  Participants are measured only with underwear cloths on the bioimpedance scale TANITA BC 602
Change in the baseline of the cardiovascular risk index with the waist-hip measurement | From enrollment to end of treatment, 9 months
  The waist-to-hip ratio (WHR) is used to estimate intra-abdominal fat and assess cardiovascular risk. It's calculated by dividing waist circumference by hip circumference (in centimetres). According to WHO, a WHR ≤ 0.80 in women and ≤ 0.95 in men indicates low risk. Moderate risk is defined as 0.81-0.85 in women and 0.96-1.00 in men. Values ≥ 0.86 in women and ≥ 1.01 in men suggest high cardiovascular risk.
Change in the baseline of food consumption frequency on 30 points of food consumption frequency questionnaire | From enrollment to end of treatment, 9 months
  The following questionnaire is to be completed by the subject in order to ascertain their habitual dietary intake. The questionnaire under consideration consists of 30 items, which have been classified into the following food groups: carbohydrates, proteins, fats, sugars, dairy products and legumes. For each item, respondents are required to indicate whether the food or drink is consumed daily, weekly, monthly, annually, or never.
Number of participants presenting abnormal laboratory results related to lipid profile. | From enrollment to end of treatment, 9 months
  In relation to the lipid profile, the following are assessed: total cholesterol, LDL, HDL and triglyceride levels mesured in mg/dL of blood.
Number of participants presenting abnormal laboratory results related to hormone levels. | From enrollment to end of treatment, 9 months
  Hormonal profile assessment includes TSH (mesured in IU/ml) and cortisol (mesured in mg/dl)
Number of participants presenting abnormal laboratory results related to liver function. | From enrollment to end of treatment, 9 months
  The hepatic profile is assessed by measuring creatinine and urea in mg/dl.
Number of participants presenting abnormal laboratory results related to blood glucose level. | From enrollment to end of treatment, 9 months
  Glucose and glycosylated haemoglobin (only in diabetic individuals) are measured in mg/dL.
Number of participants with abnormal laboratory results related to red and white blood cell series, including monocytes, leukocytes, and hematocrit. | From enrollment to end of treatment, 9 months
  Monocytes and leukocytes will be measured in ×10³/μL, and hematocrit will be expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Prats-Arimon, PHD, Principal Investigator — University of Barcelona
Locations (1):
- Agrupació Europea de Cooperació Territorial, Puigcerdà, Girona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD when the periode of collecting data is finished.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From juin 2025 until the article will be published
Access Criteria: All team researchers from University of Barcelona and Hospital de Cerdanya can share IPD throught SPSS program by corporative mail.All researchers need a password to access the institution's intranet. In addition, a shared folder will be generated where only researchers have access to share other documents

REFERENCES:
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Màs-Alòs, S., Galindo-Ortego, G., Panas-Anzano, A., Peirau-Terés, X., Real, J.(2017).Promoció de la salut i prescripció d'exercici físic des de centres d'atenció primària. Justificació i disseny. Apunts. Educació Física i Esports, 3, 40-57.
- [Background] WHO. (2015). Physical activity strategy forthe WHO European Region 2016-2025. Physical activity strategy forthe WHO European Region 2016-2025. Regional Committee for Europe 65th session (págs. 5-27). Vilnius, Lithuania: World Health Organization.
- [Background] WHO. (2013). Global action plan for the prevention and control of noncommunicable diseases 2013-2020.Geneva: World Health Organization. Obtenido de World Health Organization: (http://www.who.int/nmh/publications/ncd-action-plan/en/)
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Mollard P, Klimis S, Berard J. [Intermittent bladder catheterization many times a day. Treatment of neurogenic bladder in children]. Chir Pediatr. 1980;21(2):149-53. No abstract available. French. PMID 7448983
- [Background] Budreviciute A, Damiati S, Sabir DK, Onder K, Schuller-Goetzburg P, Plakys G, Katileviciute A, Khoja S, Kodzius R. Management and Prevention Strategies for Non-communicable Diseases (NCDs) and Their Risk Factors. Front Public Health. 2020 Nov 26;8:574111. doi: 10.3389/fpubh.2020.574111. eCollection 2020. PMID 33324597
- [Background] Celis-Morales CA, Lyall DM, Anderson J, Iliodromiti S, Fan Y, Ntuk UE, Mackay DF, Pell JP, Sattar N, Gill JM. The association between physical activity and risk of mortality is modulated by grip strength and cardiorespiratory fitness: evidence from 498 135 UK-Biobank participants. Eur Heart J. 2017 Jan 7;38(2):116-122. doi: 10.1093/eurheartj/ehw249. PMID 28158566
- [Background] Ministerio de Sanidad Consumo y Bienestar. Encuesta Nacional de Salud España 2017. Resumen Metodológico. Encuesta Nac Salud España 2017 Resum Metod. 2017; [aprox. 3 p.]. Available online: https://www.sanidad.gob.es/estadEstudios/estadisticas/ encuestaNacional/encuesta2017.htm
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Zubin Maslov P, Schulman A, Lavie CJ, Narula J. Personalized exercise dose prescription. Eur Heart J. 2018 Jul 1;39(25):2346-2355. doi: 10.1093/eurheartj/ehx686. PMID 29301027
- [Background] Liu Y, Yan T, Chu JM, Chen Y, Dunnett S, Ho YS, Wong GT, Chang RC. The beneficial effects of physical exercise in the brain and related pathophysiological mechanisms in neurodegenerative diseases. Lab Invest. 2019 Jul;99(7):943-957. doi: 10.1038/s41374-019-0232-y. Epub 2019 Feb 26. PMID 30808929
- [Background] Poon ET, Little JP, Sit CH, Wong SH. The effect of low-volume high-intensity interval training on cardiometabolic health and psychological responses in overweight/obese middle-aged men. J Sports Sci. 2020 Sep;38(17):1997-2004. doi: 10.1080/02640414.2020.1766178. Epub 2020 Jun 4. PMID 32497454
- [Background] Prats-Arimon M, Puig-Llobet M, Barcelo-Peiro O, Ribot-Domenech I, Vilalta-Sererols C, Fontecha-Valero B, Heras-Ojeda M, Aguera Z, Lluch-Canut T, Moreno-Poyato A, Moreno-Arroyo MC. An Interdisciplinary Intervention Based on Prescription of Physical Activity, Diet, and Positive Mental Health to Promote Healthy Lifestyle in Patients with Obesity: A Randomized Control Trial. Nutrients. 2024 Aug 20;16(16):2776. doi: 10.3390/nu16162776. PMID 39203911
- [Background] Brorsson Lundqvist E, Praetorius Bjork M, Bernhardsson S. Physical activity on prescription in Swedish primary care: a survey on use, views, and implementation determinants amongst general practitioners. Scand J Prim Health Care. 2024 Mar;42(1):61-71. doi: 10.1080/02813432.2023.2288126. Epub 2024 Feb 7. PMID 38047631